CLINICAL TRIAL: NCT00778960
Title: Mechanistic Pathways of Mindfulness Meditation in Post-traumatic Stress Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, Helane Wahbeh, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01AT004951-01 (NIH); K01AT004951-01 (NIH); 4692
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Post-Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Slow Breathing Group (Experimental)
  Interventions: Behavioral: Slow Breathing
- Meditation Group (Experimental)
  Interventions: Behavioral: Meditation
- Meditation and Slow Breathing Group (Experimental)
  Interventions: Behavioral: Meditation and slow breathing
- Sitting Quietly Group (Placebo Comparator)
  Interventions: Behavioral: Sitting Quietly

INTERVENTIONS:
Behavioral: Slow Breathing — The slowed breathing group will be trained on a breathing device, RESPeRATE, designed to reduce respiratory rate.They will practice with RESPeRATE once a week (for 6 weeks) in the laboratory with the research staff.
  Arms: Slow Breathing Group
Behavioral: Meditation — The Mindfulness Body Scan meditation will be used for the mindfulness meditation group.Participants will be trained once a week (for six weeks) in the laboratory by the research staff.
  Arms: Meditation Group
Behavioral: Meditation and slow breathing — A structured Mindfulness breathing will be guided by the research staff during the lab trainings. The participant will sit upright and attempt to focus attention on his or her own breath as it passes the opening of the nostrils or on the rising and falling of the abdomen or chest. Whenever attention wanders from the breath, the participant will simply notice the distracting thought and then let it go as attention is returned to the breath. Training will be given once every week for 6 weeks.
  Arms: Meditation and Slow Breathing Group
Behavioral: Sitting Quietly — The SQ control group's "intervention" will include sitting quietly and listening to a neutral-content book on tape to serve as a time and attention control at each laboratory session. They will also be asked to sit quietly at home daily.
  Arms: Sitting Quietly Group

SUMMARY:
The purpose of this study is to find out how meditation influences certain systems in the body: nervous system, hormonal system, and respiratory system. Another purpose is to see how meditation may help improve post-traumatic stress disorder symptoms.

DETAILED DESCRIPTION:
This study requires nine visits to the clinic: one screening visit, one baseline visit, six training sessions, and one endpoint visit. There will be approximately 100 people enrolled in this study who will be randomly allocated to one of four groups: a slow breathing group, a meditation group, a meditation plus slow breathing group and a sitting quietly group.

Participants will undergo a telephone screening, a screening visit, baseline visit, six intervention visits (once per week for six weeks), and one endpoint visit (one week after the final training visit). A telephone screening and screening visit will ensure participant eligibility. The screening visit included structured clinician interviews on PTSD symptoms and other mental health disorders, completion of questionnaires, and receipt of home saliva collection kit. At the baseline visit, electrodes will be attached to measure the electrical activity of head, chest, skin, and respiration and blood pressure during a computer task. Intervention visits include slow breathing, meditation, mediation and slow breathing, or sitting quietly depending on which group the participant is allocated to. Breathing rates and other electrical activity of the body will be measured also. Breathing rate will be measured with an elastic band that is placed around the chest. Electrical activity will be measured by the electrodes that will be placed on the scalp, chest and skin. The endpoint visit will be exactly the same as the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Combat veteran (defined by a score of ≥7 on the Combat exposure scale)
* Chronic PTSD diagnosis
* Age range (25-65 years)
* Both genders
* Good general medical health
* Stable dose of medications for concurrent stable medical conditions for at least 4 weeks prior to start of the study.
* Willing and able to provide informed consent.

Exclusion Criteria:

Significant chronic medical illness including:

* current cancer treatment,
* unstable angina,
* recent myocardial infarction,
* current or past history of stroke,
* transient ischemic attack,
* congestive heart failure,
* chronic renal or hepatic failure,
* hypothyroidism

Psychiatric or behavioral illness including:

* schizophrenia,
* schizoaffective disorder,
* bipolar disorder,
* psychotic disorder (not including transient dissociative states or flashbacks associated with PTSD re-experiencing symptoms),
* any DSM-IV cognitive disorder,
* current delirium,
* psychiatric instability or situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to the patient or others.
* Substance dependence disorder within 3 months of the study or
* current substance use other than alcohol (no more than 2 drinks/day by self-report)
* Sexual assault as primary PTSD event/s.
* Planning to move from the area in the next year.
* Prior or current meditation practice.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Attentional Network Task: conflict effect score | Change from Baseline to Endpoint visit (one week after last training visit)
Awakening cortisol values | Change from Baseline to Endpoint visit (one week after last training visit)
Post-traumatic stress disorder checklist-hyperarousal score | Change from Baseline to Endpoint visit (one week after last training visit)

SECONDARY OUTCOMES:
Intrusive Thought Scale | Change from Baseline to Endpoint visit (one week after last training visit)
EEG event-related negativity during Attentional Network Task | Change from Baseline to Endpoint visit (one week after last training visit)
Heart rate | Change from Baseline to Endpoint visit (one week after last training visit)

CONTACTS AND LOCATIONS:
Overall Officials: Helane Wahbeh, ND, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States